CLINICAL TRIAL: NCT00743015
Title: Relative Bioavailability Following Single Oral Administration of 200 mg of BI 44370 During and Between Migraine Attacks in Male and Female Migraine Patients. An Open-label, Fixed-sequence, Two-period Study With Intraindividual Comparison
Brief Title: Relative Bioavailability of a Single Dose of BI 44370 Tablet During and Between Migraine Attacks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Crossover | Purpose: Treatment
Other Study IDs: 1246.21; EudraCT 2008-001356-42
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

INTERVENTIONS:
Drug: BI 44370 TA tablet

SUMMARY:
The general aim is to evaluate the relative oral bioavailability of BI 44370 TA tablets during and between migraine attacks as well as Safety, Tolerability and Pharmacokinetic

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female migraine patients (age 18 to 65 years) with or without aura, diagnosed according to IHS criteria.
* Established migraine diagnosis for >= 1 year.
* Age at migraine onset <= 50 years.
* Well documented (for >= 3 months) retrospective history of migraine with headache of moderate to severe intensity and with an attack duration of at least 6 hours and migraine frequency of 2-8 times / month
* Other forms of headache are permitted if they on average occur on not more than 10 days / month and if the patient is able to differentiate migraine headache from other forms of headache.
* Patient has provided written informed consent in accordance with ICH-GCP and local legislation.
* Patient is in general good health based om screening assessment

Exclusion Criteria:

* Women of child-bearing potential without an adequate method of contraception
* Any woman of child-bearing potential not having a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline
* Breastfeeding women
* Males not willing to use adequate contraception (condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilization, IUD [intrauterine device]) during the whole study period from the time of the first intake of study drug until three months after the last intake.
* History of hemiplegic, ophthalmoplegic, or basilar migraine or cluster headache.
* History of treatment resistant migraine attacks, defined as a lack of response to a range of commonly used acute anti-migraine compounds.
* History of , clinical evidence for, or screening/baseline findings suggestive of significant medical disorders (e.g. cardiovascular, peripheral vascular, hepatic, respiratory, haematological, renal, gastrointestinal, immunological, metabolic, hormonal, neurological or psychiatric disorders)
* Smokers ... (cont.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum concentration of BI 44370 BS in plasma) | 48 hours
AUC0-2 (area under the concentration-time curve of BI 44370 BS in plasma over the time interval from 0 to 2 h after drug administration) | 48 hours
AUC0-∞ (area under the concentration-time curve of BI 44370 BS in plasma over the time interval from 0 extrapolated to infinity) | 48 hours
tmax (time from dosing to maximum measured concentration) | 48 hours

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of BI 44370 BS in plasma over the time interval from 0 to the time of the last quantifiable data point) | 48 hours
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | 48 hours
AUCt1-t2 (Area under the concentration-time curve of BI 44370 BS in plasma over the time interval t1 to t2) | 48 hours
λz (terminal rate constant in plasma) | 48 hours
t1/2 (terminal half-life of BI 44370 BS in plasma) | 48 hours
MRTp.o. (mean residence time of BI 44370 BS in the body after p.o. administration) | 48 hours
CL/F (Apparent clearance of BI 44370 BS in plasma after extravascular administration) | 48 hours
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | 48 hours
Ae0-12 (amount of BI 44370 BS eliminated in urine from time point 0 - 12 h after drug administration) | 48 hours
fe0-12 (fraction of BI 44370 BS eliminated in urine from time point 0 - 12 h after drug administration) | 48 hours
CLR,0-12 (renal clearance of BI 44370 BS from time point 0 - 12 h after drug administration) | 48 hours
Changes from baseline in Physical examination | 48 hours
Changes from baseline in Vital signs: Blood pressure (BP) and pulse rate (PR) | 48 hours
Changes from baseline in 12-lead electrocardiogram (ECG) | 48 hours
Occurrence of Adverse events (AEs) | 48 hours
Assessment of tolerability by investigator | 48 hours
Number of participants with abnormalities in clinical laboratory parameters | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- 1246.21.32001 Boehringer Ingelheim Investigational Site, Leuven, Belgium
- 1246.21.49001 Boehringer Ingelheim Investigational Site, Berlin, Germany